CLINICAL TRIAL: NCT07256652
Title: How Does YES Bar Affect Blood Glucose Levels?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 38611
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Blood Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Other: YES Bar

INTERVENTIONS:
Other: YES Bar — The YES Bar, a gluten-free, plant-based snack, has gained attention for not spiking blood glucose levels like a lot of quick packaged snack bars. An individual in the study will be provided with a mix of 6 different flavors of Yes Bar (all with generally the same ingredients and nutritional macros) and asked to conduct four individual experiments (with optional up to 6) in which they will test their blood glucose initially after fasting for two hours. Then at 15 to 30 minute intervals over the following two hours.

SUMMARY:
Curious to see if there is a sweet treat that doesn't spike your blood sugar (avoiding the energy crash, inflammation, and weight gain)? This study uses the Abbott Lingo CGM to see how your blood glucose levels responds to YES Bar-an all natural, gluten-free, plant-based bar that tastes like dessert. You'll track your levels before and after eating it to see if it fits into your metabolic health. (iOS Only)

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to rigorously evaluate the impact of Yes Bar on blood sugar levels in a real-world setting, utilizing the latest in continuous glucose monitoring technology provided by Abbott's Lingo CGM. The founder of Yes Bar initiated this study in response to numerous anecdotal reports suggesting that Yes Bar does not cause the blood sugar spikes typically associated with snack consumption. The objective is to move beyond these anecdotal experiences to gather solid, data-driven evidence regarding the metabolic effects of consuming Yes Bar.

Participants in this study will engage in a unique and personal exploration of their metabolic health by tracking their blood sugar levels in response to consuming Yes Bars. Utilizing the Abbott Lingo CGM, which currently is compatible only with the iPhone, participants will monitor their blood glucose response, enabling an individualized assessment of how Yes Bar integrates into their dietary habits and metabolic health.

This study is not solely for the purpose of marketing Yes Bars but aims to contribute valuable insights for participants themselves, providing them with concrete data on how their bodies respond to Yes Bars. By participating in at least four individual experiments with Yes Bar over a period of 7 days, participants will not only contribute to a broader understanding of the snack's metabolic impact but will also receive a $17 gift card as a token of appreciation for their contribution to this scientific inquiry.

The primary goal of this trial is to scientifically assess the blood sugar response following the consumption of Yes Bar, leveraging the capabilities of the Abbott Lingo CGM. This endeavor also seeks to evaluate the feasibility of using consumer-grade continuous blood glucose monitors in dietary impact studies, in collaboration with Efforia. Through this study, we aim to bridge the gap between anecdotal evidence and empirical data, potentially transforming the way Yes Bar is marketed and perceived in the context of a healthy diet.

This study is not only pivotal for marketing strategies but, more importantly, serves as an opportunity for participants to gain insights into their own metabolic health, offering a personalized perspective on how Yes Bar might help in avoiding the undesirable blood sugar fluctuations that lead to energy crashes and cravings. Participants will emerge from this study with personalized data that could inform their dietary choices and perhaps introduce them to a new, metabolically friendly snack option.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
After Food Glucose Follow Up | Change from baseline (Day 1-0) in blood glucose levels immediately after consuming a specific food (Day 1)
  Timed Blood Glucose Monitoring for a Specific Food is an invaluable tool for understanding individual metabolic responses to food intake. This survey involves using a continuous glucose monitor (CGM) to record blood glucose levels after consuming a specific food, helping to pinpoint how different foods impact blood sugar levels over a certain period. The data collected can significantly aid in optimizing dietary choices by demonstrating the foods that cause glucose spikes or maintain stability. Ultimately, the insights gained can lead to improved metabolic health, better energy levels, and an enhanced overall well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=38611